CLINICAL TRIAL: NCT01474603
Title: IMpact of n-3 Polyunsaturated Fatty Acids With a Protein-Enriched DiEt With Low Glycemic Index on Metabolic and Inflammatory Parameters in Type 2 Diabetic and Obese Patients: an Observational Pilot Study
Brief Title: Impact of n-3 Polyunsaturated Fatty Acids in a Protein-enriched Diet With Low GI in Type 2 Diabetes Patients
Acronym: IMPEDE-DM2
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Enervit Spa (company) (Unknown)
Responsible Party: Principal Investigator, Thomas M Stulnig, Associate Professor, Medical University of Vienna
Other Study IDs: IMPEDE-DM2
Record Dates: First submitted 2011-11-15; First posted 2011-11-18 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Overweight; Obese; Insulin Resistance; Diabetes
Keywords: observational study
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance; Diabetes Mellitus | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma samples for biochemical analyses
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: overweight or obese diabetic
  Interventions: Dietary Supplement: n-3 PUFA in protein-enriched low-GI diet

INTERVENTIONS:
Dietary Supplement: n-3 PUFA in protein-enriched low-GI diet — 3 g per day n-3 polyunsaturated fatty acids in a protein-enriched low-GI diet

SUMMARY:
Type 2 diabetes is tightly associated with overweight and obesity. Inflammatory processes are crucial triggers for insulin resistance that paves the way to type 2 diabetes. In a previous study the investigators have shown that n-3 polyunsaturated fatty acids diminish adipose tissue inflammation in morbidly obese non-diabetic subjects. in this observational study the investigators will apply n-3 polyunsaturated fatty acids as addition to a protein-enriched diet with low glycemic index to overweight and obese patients with insulin resistance, prediabetes and manifest type 2 diabetes over up to 6 months. Primary efficacy parameters are changes from baseline in HbA1c and body weight for for type 2 diabetes and all other patients, respectively.

ELIGIBILITY:
Inclusion Criteria:

* overweight or obesity AND
* insulin resistant OR pre-diabetes OR type 2 diabetes

Exclusion Criteria:

* changes in anti-diabetic medication in the lat two months
* acute illness during the last two weeks
* HIV infection
* hepatitis of other clinically significant hepatic disease other than non-alcoholic hepatic steatosis
* severe or insufficiently treated cardiovascular, renal (GFR-MDRD < 60 ml/min) or pulmonary disease
* Macroproteinuria (> 300 mg/g creatinine)
* clinically significant or insufficiently treated thyroid disease
* anemia
* active malignant disease
* inborn or acquired coagulopathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: overweight to obese insulin resistant, prediabetic and diabetic patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2014-11 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
HbA1c change from baseline (type 2 diabetes patients) | 3 months
body weight change from baseline (non-diabetic patients) | 3 months

SECONDARY OUTCOMES:
change from baseline of inflammatory and metabolic parameters | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. Medicine III, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Moosheer SM, Waldschutz W, Itariu BK, Brath H, Stulnig TM. A protein-enriched low glycemic index diet with omega-3 polyunsaturated fatty acid supplementation exerts beneficial effects on metabolic control in type 2 diabetes. Prim Care Diabetes. 2014 Dec;8(4):308-14. doi: 10.1016/j.pcd.2014.02.004. Epub 2014 Mar 19. PMID 24656509